CLINICAL TRIAL: NCT02192697
Title: An Open-label Study of the Oral Administration of ASP8273 in Patients With Non-small Cell Lung Cancer Harboring Epidermal Growth Factor Receptor (EGFR) Mutations
Brief Title: An Open Study of ASP8273 in Patients With Non-Small-Cell Lung Cancer (NSCLC) Who Have Epidermal Growth Factor Receptor (EGFR) Mutations
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Following recommendation by SOLAR Study IDMC, Astellas closed enrollment in ASP8273 studies.
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8273-CL-0101
Record Dates: First submitted 2014-05-28; First posted 2014-07-17 (Estimated); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Non-small Cell Lung Cancer
Keywords: safety; pharmacokinetics; tolerability; ASP8273; Non-small Cell Lung Cancer; T790M resistance mutation; NSCLC; Epidermal Growth Factor Receptor mutations; irreversible EGFR inhibitor; antitumor activity; EGFR
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — naquotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Phase I dose-escalation group (Experimental): Oral administration
  Interventions: Drug: ASP8273
- Phase I EGFR-T790M mutation group (Experimental): Oral administration
  Interventions: Drug: ASP8273
- Phase II group (Experimental): Oral administration
  Interventions: Drug: ASP8273

INTERVENTIONS:
Drug: ASP8273 — Oral administration

SUMMARY:
Purpose of the study is to determine the following in patients with non-small cell lung cancer (NSCLC) harboring EGFR activating mutations.

* the safety and tolerability of ASP8273.
* the pharmacokinetics (PK) of ASP8273.
* the antitumor activity of ASP8273.

DETAILED DESCRIPTION:
This study consists of Phase I and Phase II.

The objectives of Phase I are to determine the following in patients with non-small cell lung cancer (NSCLC) harboring EGFR activating mutations.

* safety and tolerability of ASP8273.
* the maximum tolerated dose (MTD) and/or recommended phase II dose (RP2D) of ASP8273 based on the dose limiting toxicity (DLT) profile.
* pharmacokinetics (PK) of ASP8273.
* antitumor activity of ASP8273.

The objectives of Phase II are to determine the following at the RP2D of ASP8273 in patients with NSCLC harboring EGFR mutation.

* efficacy of ASP8273
* safety of ASP8273
* PK of ASP8273

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of NSCLC.
* Patients confirmed to have the del ex19, L858R, G719X, or L861Q mutation among the EGFR activating mutations (patients at the study site who are documented to have any of the above-stated EGFR activating mutations can be enrolled in the study).
* Life expectancy ≥ 12 weeks based on the investigator's/subinvestigator's judgment.
* [Phase I]

  * Patients who have previously been treated with EGFR tyrosine-kinase inhibitors (EGFR-TKIs)*
  * Those who are not expected to show a therapeutic response to existing treatments in the investigator's/subinvestigator's opinion.
* [Phase II]

  * Patients who have been confirmed to have progressive disease (PD) after previous treatment with EGFR-TKIs*; for those who have received 2 or more regimens of previous treatment, the last regimen before enrollment should have included EGFR-TKIs.
  * *Erlotinib, gefitinib, and EGFR-TKIs under clinical investigation (e.g., neratinib, afatinib, dacomitinib)
  * Expression of the EGFR-T790M mutation as confirmed by a tumor biopsy of the primary or metastatic lesions after confirmation of PD following previous treatment with EGFR-TKIs and before enrollment, or by a tumor tissue sample that had been collected and archived after confirmation of PD following previous treatment with EGFR-TKIs.
  * At least 1 measurable lesion based on Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.

Exclusion Criteria:

* Persistent clinical evidence of previous antitumor treatment related toxicity ≥ Grade 2 using the Japan Clinical Oncology Group (JCOG) Japanese translation of the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 (NCI CTCAE v4.0 - JCOG) (except alopecia and skin toxicities considered irrelevant in study enrollment by the investigator/sub-investigator).
* History of or concurrent interstitial lung disease
* Received treatment with a reversible EGFR-TKI (erlotinib or gefitinib) within 8 days before the start of the study treatment.
* Received previous treatment (except reversible EGFR-TKIs) intended to have antitumor effects or treatment with another investigational drug or an investigational device within 14 days before the start of the study treatment.
* Previously received treatment with EGFR-TKIs (e.g., CO-1686, AZD9291) that can inhibit EGFR with the T790M mutation.
* It is planned that the subject will undergo a surgical procedure during the course of the study or the subject still has an unhealed wound after previous surgery
* Symptomatic central nervous system (CNS) lesions.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2014-01-23 (Actual); Primary Completion 2016-01-15 (Actual); Study Completion 2017-06-14 (Actual)

PRIMARY OUTCOMES:
Phase I: Safety and tolerability of ASP8273 as assessed by Dose Limiting Toxicities (DLTs) | Up to Day 23
  A DLT is defined as any pre-determined toxicity that is related to study drug per the investigator and which occurs during Cycle 0 and Cycle 1 using the Japan Clinical Oncology Group (JCOG) Japanese translation of the Common Terminology Criteria for Adverse Events version 4.0 (CTCAE ver 4.0 - JCOG)
Phase II: Overall response rate (CR+PR) at Week 24 | Week 24
  The overall response rate, which is defined as the proportion of subjects whose best overall response is rated as complete response (CR) or partial response (PR) according to RECIST Version 1.1, will be calculated

SECONDARY OUTCOMES:
Phase I: Safety and tolerability of ASP8273 as assessed by adverse events (AEs) | Up to 18 months
  An AE is defined as any untoward medical occurrence in a subject administered a study drug or has undergone study procedures and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product
Phase I: Safety and tolerability of ASP8273 as assessed by laboratory tests | Up to 18 months
  Laboratory tests to be conducted are hematology, biochemistry, urinalysis, coagulation profile, lipid panel and lymphocyte subpopulation
Phase I: Safety and tolerability of ASP8273 as assessed by vital signs | Up to 18 months
  Vital signs to be measured includes blood pressure, pulse rate and temperature
Phase I: Safety and tolerability of ASP8273 as assessed by 12-lead ECG | Up to 18 months
  including the assessment of QT intervals
Phase I: Plasma concentrations of unchanged ASP8273 | Up to Day 1 of Cycle 3
Phase I: Urine concentrations of unchanged ASP8273 | Up to Day 1 of Cycle 3
Phase I: Overall response rate (CR+PR) | Up to 18 months
  The overall response rate is defined as the proportion of subjects whose best overall response is rated as complete response (CR) or partial response (PR) according to RECIST Version 1.1, will be calculated
Phase I: Disease control rate (CR+PR+SD) | Up to 18 months
  The disease control rate is defined as the proportion of subjects whose best overall response is rated as CR, PR, or stable disease (SD) according to RECIST Version 1.1, will be calculated.
Phase II: Plasma concentrations of unchanged ASP8273 | Up to Day 1 of Cycle 3
Phase II: Urine concentrations of unchanged ASP8273 | Up to Day 1 of Cycle 3
Phase II: Safety and tolerability of ASP8273 as assessed by adverse events (AEs) | Up to 18 months
  An AE is defined as any untoward medical occurrence in a subject administered a study drug or has undergone study procedures and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product
Phase II: Safety and tolerability of ASP8273 as assessed by laboratory tests | Up to 18 months
  Laboratory tests to be conducted are hematology, biochemistry, urinalysis, coagulation profile, lipid panel and lymphocyte subpopulation
Phase II: Safety and tolerability of ASP8273 as assessed by vital signs | Up to 18 months
  Vital signs to be measured includes blood pressure, pulse rate and temperature
Phase II: Safety and tolerability of ASP8273 as assessed by 12-lead ECG | Up to 18 months
  including the assessment of QT intervals
Phase II: Disease control rate | Up to 18 months
  The disease control rate is defined as the proportion of subjects whose best overall response is rated as CR, PR, or stable disease (SD) according to RECIST Version 1.1, will be calculated.
Phase II: Progression-free survival (PFS) | Up to 18 months
Phase II: Overall survival (OS) | Up to 18 months
Phase II: Overall response rate (CR+PR) | Up to 18 months
  The overall response rate, which is defined as the proportion of subjects whose best overall response is rated as complete response (CR) or partial response (PR) according to RECIST Version 1.1, will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (14):
- Japan (9):
  - Site: 4, Fukuoka
  - Site: 9, Fukuoka
  - Site: 8, Miyagi
  - Site: 7, Okayama
  - Site: 3, Osaka
  - Site: 6, Osaka
  - Site: 2, Shizuoka
  - Site: 1, Tokyo
  - Site: 5, Tokyo
- South Korea (3):
  - Site: 10, Seoul
  - Site: 11, Seoul
  - Site: 12, Seoul
- Taiwan (2):
  - Site: 13, Taipei
  - Site: 14, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=259